CLINICAL TRIAL: NCT01375868
Title: Phase IIIb Study of Recombinant Tetravalent HPV Vaccine in Patients With Recurrent Respiratory Papillomatosis
Brief Title: Effect of Vaccination in Patients With Recurrent Respiratory Papillomatosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ruth Tachezy, PhD. (Other)
Collaborators: Medical Healthcom Prague (Unknown); Na Homolce Hospital (Other)
Responsible Party: Sponsor-Investigator, Ruth Tachezy, PhD., M.Sc., PhD., Institute of Hematology and Blood Transfusion, Czech Republic
Organization: Institute of Hematology and Blood Transfusion, Czech Republic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHKT-RLP/2011; 2011-002667-14 (EudraCT Number)
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Squamous Papilloma of the Larynx
Keywords: HPV; recurrent respiratory papillomatosis; antibodies
MeSH Terms: conditions — Laryngeal papillomatosis; Recurrent respiratory papillomatosis | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vaccine Silgard (Experimental): vaccination with tetravalent antiviral vaccine, 3 doses
  Interventions: Biological: Silgard

INTERVENTIONS:
Biological: Silgard — vaccination with tetravalent antiviral vaccine

SUMMARY:
Vaccines against human papillomaviruses are now commercially available. One of the commercial vaccine contains antigens of both LR HPV types which cause virtually all cases of RRP. Clinical trials have documented the safety and immunogenicity of this vaccine as well as its effectiveness in prevention of incident and persistent infection of the vaccinal types as well as a development of lesions caused by these types. After vaccination the antibodies level increases dramatically and the high levels of antibodies are present in the blood still after 6 years. Furthermore, the neutralization antibodies to the vaccinal antigens have been detected in the cervical mucus of vaccinated women. The preliminary data are now available showing the presence of HPV-specific antibodies in the oral cavity in women after vaccination. The level of antibodies has been dependent on time since vaccination.

DETAILED DESCRIPTION:
In our previous studies we have documented that in patients with RRP the level of HPV-specific antibodies is low and increases only after numerous surgery procedures. Therefore the application of this vaccine to patients with RRP can stimulate increased level of antibodies in the blood as well as presence of virus-specific neutralization antibodies on the surface of upper aero digestive tract and neutralize viruses shed from new papillomas and in this way protect patient from spreading of the infection as well as to facilitate the decrease of load of infectious virus shed from the lesion. This can possibly lead to the inhibition of growth of the papillomatous lesion.

ELIGIBILITY:
Inclusion Criteria:

Patients with RRP which sign the informed consent form with both parts of the study will be enrolled.

Exclusion Criteria:

Patients who experience severe side effects of vaccination after the first or second dose will not be vaccinated with the third dose and they will be excluded from the study. Patients who will not receive all three doses within one year and 30 days will be also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-10; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
occurrence or frequency of recurrences of laryngeal papillomatosis | 5 years
  The main aim is to evaluate the effect of tetravalent HPV vaccine on occurrence or frequency of recurrences of laryngeal papillomatosis.

SECONDARY OUTCOMES:
HPV type present in the tissue | 2 years
  We will determine the type of human papillomavirus present in the surgically removed tissue.
the presence of HPV specific antibodies | 5 years
  We will evaluate the presence of HPV-specific antibodies in sera of patients with recurrent papillomatosis before and after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Tachezy, PhD., Principal Investigator — Institute of Hematology and Blood Transfusion
Locations (1):
- Institute of Hematology and Blood Transfusion, Prague, Czechia

REFERENCES:
- [Background] Tachezy R, Hamsikova E, Valvoda J, Van Ranst M, Betka J, Burk RD, Vonka V. Antibody response to a synthetic peptide derived from the human papillomavirus type 6/11 L2 protein in recurrent respiratory papillomatosis: correlation between Southern blot hybridization, polymerase chain reaction, and serology. J Med Virol. 1994 Jan;42(1):52-9. doi: 10.1002/jmv.1890420111. PMID 8308521
- [Derived] Smahelova J, Hamsikova E, Ludvikova V, Vydrova J, Traboulsi J, Vencalek O, Lukes P, Tachezy R. Outcomes After Human Papillomavirus Vaccination in Patients With Recurrent Respiratory Papillomatosis: A Nonrandomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2022 Jul 1;148(7):654-661. doi: 10.1001/jamaoto.2022.1190. PMID 35653138